CLINICAL TRIAL: NCT00860600
Title: The Clinical Trial of PG2 in Subjects With Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: Safety and Efficacy Study of PG2 to Treat Idiopathic Thrombocytopenic Purpura (ITP) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-CP014
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Thrombocytopenic Purpura (ITP)
Keywords: Idiopathic Thrombocytopenic Purpura (ITP); Platelet Response; PG2 Treatment; Quality of Life; Fatigue; WHO Bleeding score
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. PG2 Treatment: 5 days/week (Experimental): Powder for Injection, 500 mg PG2/500 ml normal saline, 5 days/week, 2 to 4 weeks
  Interventions: Drug: PG2
- 2. PG2 Treatment: 3 days/week (Experimental): Powder for Injection, 500 mg PG2/500 ml normal saline, 3 days/week, 2 to 4 weeks
  Interventions: Drug: PG2

INTERVENTIONS:
Drug: PG2 — 500mg/vial, iv infusion, 3 ~ 5 times/week, 2.5 ~ 3.5 hr/time
  Other Names: PG2 Injection 500 mg

SUMMARY:
This was a phase II multi-center, randomized, open-label study with two parallel study groups to evaluate the efficacy and safety of PG2 in ITP patients.

DETAILED DESCRIPTION:
The primary objective of this exploratory study is to evaluate the efficacy of PG2 in raising the platelet counts in ITP patients using two dosing schedules. The secondary objective is to determine the safety of PG2 treatment among these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Confirmed diagnosis of chronic ITP, according to The American Society of Hematology (ASH) Guidelines, for at least 6 months and have received one or more prior conventional treatments for ITP.
3. Patient's platelet count of less than 50,000 per cubic millimeter at enrollment, platelet count is calculated from the mean of 2 platelet counts taken during the screening period and that on day1.
4. The subject or his/her legal delegate has signed an informed consent form.
5. Absence of other conditions that, in the opinion of the investigator, could cause thrombocytopenia.
6. If subjects are currently being treated with corticosteroids, the treatment regimen/dose must have been stable (±25% total dose/day) for a minimum of 4 weeks before screening. However, subjects must remain on a stable treatment regimen. If there is any intent to alter the corticosteroid treatment regimen (e.g., tapering of corticosteroids) before Day 10, subjects may not be included in the study.
7. If subjects are currently being treated with cyclophosphamide, azathioprine or attenuated androgens, the treatment regimen and dose must have been stable (±25% total dose/day) for a minimum of 3 months before screening. However, if there is any intent to alter the treatment regimen before Day 10, subjects may not be included in the study.
8. If a subject is a female of child-bearing potential, she must have a negative result on a urine-based HCG pregnancy test.
9. If a subject is of child-bearing potential, he/she must practice contraception by using a method of proven reliability for the duration of the study.

Exclusion Criteria:

1. The subject has a history of any severe or anaphylactic reaction to blood or any blood-derived product, or any severe reaction to IVIG or any other IgG preparation.
2. The subject is known to be intolerant to any component of the investigational product.
3. The subject has received any live virus vaccine within the last 3 months.
4. The subject has received an IVIG preparation within 1 month prior to screening.
5. The subject is currently receiving, or has received, any investigational agent within one month prior to screening.
6. The subject has received Rituximab within 3 months before screening.
7. The subject is pregnant or is nursing.
8. The subject is diagnosed of having HIV.
9. The subject, at screening, has levels greater than 2.5 times the upper limit of normal liver function of alanine aminotransferase or aspartate aminotransferase.
10. The subject has a severe renal impairment (defined as serum creatinine greater than 2 times the upper limit of normal or BUN greater than 2.5 times the upper limit of normal for range); or the subject is on dialysis.
11. The subject has a history of deep vein thrombosis (DVT) or thrombotic complications.
12. The subject has any history of hyperviscosity, transient ischemic attack (TIA), stroke, other thromboembolic event, or unstable angina.
13. The subject suffers from any acute or chronic medical conditions (e.g., renal disease or predisposing conditions for renal disease, coronary artery disease, or protein losing enteropathy) that, in the opinion of the investigator, may interfere with the conduct of the study.
14. The subject has an acquired medical condition, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (defined as an absolute neutrophil count (ANC) < 1 x 109/L) or has been diagnosed as non-ITP patients.
15. The subject is unlikely to adhere to the protocol requirements of the study or is likely to be uncooperative.
16. The subject is unwilling or unable to answer the quality of life questionnaires i.e. the BFI.
17. The subject has undergone splenectomy within 4 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Platelet Response | 17 weeks

SECONDARY OUTCOMES:
The total number of bleeding events Grade 2 or higher for each subject during the treatment period, or till the time of end-of-study visit for early withdrawal patients | 17 weeks
The subject incidence of requiring rescue therapy during the treatment period | 17 weeks
The endogenous TPO and anti-platelet antibody levels | 17 weeks
Patient's fatigue status (measured by the Brief Fatigue Inventory) | 17 weeks
Patient's Bleeding Score (measured by the WHO Bleeding Scale) | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Fung Lin, M.D., Ph.D., Study Chair — E-Da Cancer Hospital
Locations (4):
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei